CLINICAL TRIAL: NCT06187415
Title: Harm Reduction Strategies for Gay, Bisexual and Other Men Who Have Sex With Men Engaging in Chemsex
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: Healing, Empowerment, Recovery of Chemsex (HERO) integrated care clinic (Unknown)
Responsible Party: Principal Investigator, Carol Strong, Associate Professor, National Cheng Kung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HarmReductionAPPService
Record Dates: First submitted 2023-11-30; First posted 2024-01-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Harm Reduction
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The harm reduction mobile app (Experimental): Participants in the intervention arm will receive access to all the app functions. The primary features of the app include PrEP taking diary, setting harm reduction goals, providing location of needle and syringe services program, providing accurate information on chemsex urban legends, and sending alerts to emergency contact in case of intoxication.
  Interventions: Behavioral: Mobile app to reduce harm of chemsex

INTERVENTIONS:
Behavioral: Mobile app to reduce harm of chemsex — Access to the mobile app which includes PrEP diary, demistification of chemsex urban legends, information on the location of needle and syringe services program, and alert sending to emergency contact.

SUMMARY:
This study is examining the usability and effectiveness of an innovative mobile app that integrates harm reduction strategies into the existing pre-exposure prophylaxis (PrEP) intake and adherence app, with an overarching goal to reduce the potentially negative consequences of problematics chemsex behavior for individuals and communities.

DETAILED DESCRIPTION:
The practice of sexualized drug use is historical and has been noted across a diversity of genders and people of various sexual orientations. The term "chemsex" has been used to specifically describe the use of psychoactive substances in sexualized settings among gay, bisexual, and other men who have sex with men (GBMSM), particularly stimulants like methamphetamine and mephedrone, or other drugs like γ-hydroxybutyrate (GHB), γ-butyrolactone (GBL). Chemsex among GBMSM has coincided with the emergence of sexual-networking mobile apps, creating new opportunities for finding new partners with the intention to engage in chemsex.

Harm reduction strategies for GBMSM engaging in chemsex are needed because the use of these drugs can have negative consequences for the physical and mental health of the people who use them. One of the main risks associated with chemsex is the possibility of overdose. In addition to the risk of overdose, chemsex may also increase the risk of sexually transmitted infections (STIs) and HIV transmission due to the higher possibility to engage in risky sexual behaviors.

Seeking help can be difficult for GBMSM who engage in chemsex due to stigma, making the harm reduction approach equally important as clinical treatment or intervention that emphasized an abstinence approach. Harm reduction strategies recognize that drug use is a complex issue and that it is not always possible or desirable for people to stop using drugs completely. Instead, harm reduction approaches aim to reduce the harm that can result from drug use and to support people in making healthier choices.

Considering also that mobile applications are another way to provide help to hard to reach population, this study aims to develop an innovative mobile app that integrates harm reduction strategies into the existing pre-exposure prophylaxis (PrEP) intake and adherence app. PrEP is a medication that can be taken daily to reduce the risk of HIV transmission. The aim of including PrEP adherence in the self-help harm reduction strategy is to ensure that participants have access to and are using an effective HIV prevention method. Behavior regulation strategies such as providing education about the risks of drug use, overdose prevention and management, and HIV prevention through correct PrEP intake, can be integrated into a mobile app that aims to minimize the negative consequences of drug use and reduce the risks associated with it, with an overarching goal to reduce the potentially negative consequences of problematics chemsex behavior for individuals and communities.

ELIGIBILITY:
Inclusion Criteria:

* individuals need to have a history of drug use (ecstasy, ketamine, crystal methamphetamine, mephedrone, and/or GHB/GBL)in a sexualized context in the previous year
* can read and understand chinese,
* willing to communicate with the research team through the mobile messenger app Line.

Exclusion criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — chemsex engaging individuals aged 18 years or older that are cisgender men or transgender female who have sex with men are eligible for the study.
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Usability of the app | 1 month
  Scores on the translated version of the mHealth App Usability questionnaire will be used to assess usability. Responses to the statements on the questionnaire ranged from 1(strongly agree) to 7 (strongly disagree). The questionnaire is the total score of each item divided by the number of items. The closer the mean value is to 1, the higher the app's usability will be.
Feasibility of the app | 1 month
  Feasibility of the app will be measured by assessing the user's frequency of app log-ins, use of app components, and duration of app use.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Strong, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- NationalCKU, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No